CLINICAL TRIAL: NCT02098330
Title: The Efficacy of Steroid Therapy in Vestibular Neuritis Confirmed by Head Impulse Test: Prospective Randomized Controlled Study
Brief Title: The Efficacy of Steroid Therapy in Vestibular Neuritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hong Ju Park, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVNHIT_kr
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Vestibular Neuritis
Keywords: Vestibular neuritis; Vertigo; Head impulse test; Steroid
MeSH Terms: conditions — Vestibular Neuronitis; Vertigo | interventions — Ginkgo Extract; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- : Ginkgo biloba & methylprednisolone (Active Comparator): Patients receive Ginkgo biloba & methylprednisolone per oral.
  Interventions: Drug: Ginkgo biloba & Methylprednisolone
- Ginkgo biloba (Placebo Comparator): Patients receive Ginkgo biloba per oral.
  Interventions: Drug: Ginkgo biloba

INTERVENTIONS:
Drug: Ginkgo biloba & Methylprednisolone — Ginkgo biloba 160 mg/day (per oral, 80 mg twice a day) for 1 month. Methylprednisolone 48 mg/day(per oral, once a day for first 9 days. And then methylprednisolone tapering was started every 2 days. The entire duration of methylprednisolone treatment was 14 days.
  Other Names: Ginexin; Methylprednisolone
  Arms: : Ginkgo biloba & methylprednisolone
Drug: Ginkgo biloba — Ginkgo biloba 160 mg/day (per oral, 80 mg twice a day) for 1 month.
  Other Names: Ginexin
  Arms: Ginkgo biloba

SUMMARY:
The purpose of this study was to compare the treatment effectiveness of steroid therapy for vestibular neuritis by using video head impulse test.

DETAILED DESCRIPTION:
This study was a prospective, randomized controlled study. The enrolled vestibular neuritis patients were randomized to conservative treatment or steroid treatment when they are diagnosed with caloric test. After initial vestibular work-up including caloric, video head impulse tests, and a questinnaire (DHI), the patient was examined with the same tests again at 6 months later. The efficacy of steroid for the patients with vestibular neuritis would be determined by the comparison of the data of each group.

ELIGIBILITY:
Inclusion Criteria:

* Ages over 18 years
* Acute vertigo that occurred within 7 days
* The spontaneous nystagmus should be detected
* Caloric weakness over 20%

Exclusion Criteria:

* Suspicious or verified a central nervous system lesion
* If the patient has denied.
* Other otologic disease (acute/chronic otitis media, otosclerosis, etc)
* The patient with history of otologic surgery
* The patient with history of brain surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The improvement in vestibular function test (caloric & videop HIT) after treatment | The first results were collected at initial diagnosis. And following results were collected 6 months after the first exam.
  The effectiveness of steroid therapy was determined by comparing the improvement of vestibular function (the degree of canal paresis by caloric test; gain and presence of refixation-saccade by video HIT test).

SECONDARY OUTCOMES:
The improvement in dizziness handicap inventory after treatment | The first results were collected at initial diagnosis. And following results were collected 6 months after the first exam.
  The effectiveness of steroid therapy was determined by comparing improvement of subjective symptoms (symptom score by DHI) in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ju Park, Professor, Study Director — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Yoo MH, Yang CJ, Kim SA, Park MJ, Ahn JH, Chung JW, Park HJ. Efficacy of steroid therapy based on symptomatic and functional improvement in patients with vestibular neuritis: a prospective randomized controlled trial. Eur Arch Otorhinolaryngol. 2017 Jun;274(6):2443-2451. doi: 10.1007/s00405-017-4556-1. Epub 2017 Apr 8. PMID 28391531